CLINICAL TRIAL: NCT05375266
Title: Immune Biomarker Study for Head and Neck Cancer
Acronym: ImmunBio-KHT
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University Hospital Erlangen (Other); University Hospital Regensburg (Other); University Hospital Augsburg (Other)
Responsible Party: Sponsor
Other Study IDs: 12-384-B
Record Dates: First submitted 2022-03-29; First posted 2022-05-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer; Oral Cavity Cancer; Oropharyngeal Cancer; Hypopharyngeal Cancer; Laryngeal Cancer
Keywords: Immunologic markers; Immunotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Cohort: The study cohort consist of patients with newly diagnosed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, paranasal sinuses or larynx in stage UICC (Union internationale contre le cancer) II-IVB
  Interventions: Other: Sampling
- Control Group: The control group consists of patients with no current diagnoses of cancer undergoing surgery at the participating medical center
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — This is an observational study. Consequently, study participation does not alter the therapy of the treated disease. Blood will be drawn from patients at several time points during and after radiotherapy (RT) and therapy with immune checkpoint inhibitor (ICI) for detailed immunomonitoring of the patients. In addition, faeces and sputum of the patients for microbiomic and metabolomic measures will be collected. Whenever possible, adequate tissue samples are taken from the center of the tumor and a biopsy is taken from the edge of the tumor including the adjacent mucosa in the nearby area without affecting the pathological assessment (study group). Blood, faeces and sputum will be taken from patients of the control group prior to surgery. After surgery, only blood will be taken.

SUMMARY:
The aim of this prospective non-interventional multi-center trial is to study the prognostic value of intratumoral and systemic immune biomarkers in newly diagnosed non-metastatic head and neck cancer. Furthermore, the local immunological processes in the tumor will be correlated with the systemic immune status determined in the peripheral blood to identify prognostic immune signatures. In addition, tumor organoids will be generated ex vivo for functional biological analyses. The main objective is to create a prognostic score determined by clusters based on tumor immunologic criteria.

DETAILED DESCRIPTION:
Except for human papillomavirus(HPV)-associated oropharyngeal cancer, immunological biomarkers do not influence treatment algorithms in locally advanced head and neck cancer. In the meantime, a prognostic significance of tumor infiltrating lymphocytes has been recognized. However, these biomarkers do not influence clinical decisions. This may be due to previous focus on the entire group of heterogeneous squamous cell carcinomas in the head and neck region, while the tumor localization has been neglected. In addition, the isolated observation of singular immune cell populations may not be sufficient with regard to the complex interactions of the tumor with the local and systemic immune system, e.g. the presence of regulatory T cells (FoxP3+) in immunologically highly active tumors ("inflamed" or "hot") improves the prognosis, whereas the prognosis is worsened in immunologically less active tumors ("immune desert").The immune checkpoint molecule programmed death-ligand 1 (PD-L1) is currently used as a single predictive marker for immunotherapy with PD(L)-1 inhibitors. Certainly, combined prospective analyses of immune cells and immune checkpoint molecules in large patient cohorts are scarce so far. Of note, the prognostic relevance of immune cells and immunologically active substances in the peripheral blood serving as makers for immunotherapies has already been described. Yet prognostic and predictive markers in the peripheral blood have rarely been studied or linked to the local tumor immune status. However, analyses of single biomarkers of local and systemic immune responses and different immune cell populations can be expected to gain prognostic precision through cluster formation and allow grouping of head and neck tumors according to immunobiological criteria rather than anatomic localization. Therefore, the investigators expect to be able to identify an immunobiological biomarker signature for head and neck tumors that will contribute to the development of future individualized treatment approaches leading to precision head and neck oncology.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, paranasal sinuses or larynx in stage UICC II-IVB (study group)
* Diseases other than malignant diseases (patients with the indication for surgery of the ear, nose nose or maxillofacial surgery) (control group)
* Absence of a currently existing or previous malignant disease regardless of the anatomical localization (control group)
* Agreement of the patients for sampling blood, saliva and stool as well as consent to the preservation of all samples for further study purposes
* Age ≥ 18 years
* Cognitive ability of the patients to understand the meaning and purpose of the study and agree to it

Exclusion Criteria:

* Distant metastases and / or simultaneous secondary carcinoma at the time of diagnosis (= inclusion date)
* Carcinomas in which it is (likely) impossible to take a sample without interfering with the further pathological assessment
* Present drug abuse
* Patients who are unable or unwilling to behave and receive treatment according to protocol
* Patients who are legally patronized
* Patients who are not eligible for participation in the study due to language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for treatment at the participating study centers and meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Observation of changes in an established immune matrix (intratumoral and systemic) of responding/non-responding patients at certain points in time in the course of treatment | Change of the immune matrix from baseline (before surgery; day0) and after surgery (day 7) and at the end of radiotherapy (day 60-70) and end of study period up to 5 years
  Based on the intrinsic immunological biology of the tumors, different immune cells and tumor cell markers will characterize immunological groups using cluster analysis.
  Immune matrix of patients assessed by LIPS (liquid immune profile-based signature) (acc. Zhou et al. JITC 2021) and Tumour Associated Lymphocytes (TAL).

SECONDARY OUTCOMES:
Longitudinal immunophenotyping of the patients: Detection of about 30 distinct immune cell (sub)types together with their activation markers during study period | The analyses are conducted at time points before (day 0) surgery and after surgery (day 7) as well as at the end of radiotherapy (day 70-80) or end of study period up to 5 years
  The distribution of immune cells and messenger substances in the blood will be examined by means of immunophenotyping in order to add the systemic immune cell composition.
  Flow cytometric assessment of the amount of circulating immune cell-distribution per milliliter whole blood according to the LIPS (liquid immune profile-based signature) technique (Zhou et al. JITC 2021).
Analysis of cytokines in peripheral blood and their change at certain points in the course of treatment | The analyses are conducted at time points before (day 0) surgery and after surgery (day 7) as well as at the end of radiotherapy (day 70-80) or end of study period up to 5 years
  Electrochemiluminescent MULTI-ARRAY measurement of concentration (pg/ml whole blood) cytokines/chemoattractant cytokines in the serum/plasma of the patients according to the LIPS (liquid immune profile-based signature) technique (Zhou et al. JITC 2021).
Determination of transcription processes in the immune cells at certain points in the course of treatment to extend the prognostic immune signature | The analyses are conducted at time points before (day 0) surgery and after Surgery (day 7) as well as at the end of radiotherapy (day 70-80) or end of study period up to 5 years
  Genetic profiling (Whole exome sequencing, RNASeq, ddPCR, realtimePCR) of transcribed genes in blood lymphocytes.
Analysis of patient's metabolic state | The analyses are conducted at time points before (day 0) surgery and after Surgery (day 7) as well as at the end of radiotherapy (day 70-80) or end of study period up to 5 years
  Massspectometric untargeted metabolomic of patients serum/plasma to assess the change of metabolites (pg/ml whole blood) from baseline to end of radiotherapy.
Analysis of patient's microbiomic state by examination of saliva, tumor and stool | The analyses are conducted at time point before surgery (day 0)
  16S rRNA deep sequencing of microbiome in salvia, tumour and stool samples to assess the presence and relative distribution of microbiotes (Operational taxonomic units [OTUs]).

CONTACTS AND LOCATIONS:
Overall Officials: Antoniu-Oreste Gostian, PD Dr. med., Study Director — ENT - Head and Neck Surgery Department, University of Erlangen-Nurnberg; Markus Hecht, PD Dr. med., Study Director — Radiation Oncology, University of Erlangen-Nurnberg; Manuel Weber, PD Dr. med. Dr. med. dent., Principal Investigator — Maxillo-facial-surgery, University of Erlangen-Nurnberg; Udo Gaipl, Prof. Dr. rer. nat. habil., Principal Investigator — Translational Radiobiology, University of Erlangen-Nurnberg; Benjamin Frey, PD Dr.-Ing. Dr. habil. med., Principal Investigator — Translational Radiobiology, University of Erlangen-Nurnberg
Locations (3):
- Germany (3):
  - ENT - Head and Neck Surgery Department, Erlangen, Bavaria
  - Maxillo-Facial-Surgery Department, Erlangen, Bavaria
  - Radiation Oncology Department, Erlangen, Bavaria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] O'Sullivan B, Huang SH, Su J, Garden AS, Sturgis EM, Dahlstrom K, Lee N, Riaz N, Pei X, Koyfman SA, Adelstein D, Burkey BB, Friborg J, Kristensen CA, Gothelf AB, Hoebers F, Kremer B, Speel EJ, Bowles DW, Raben D, Karam SD, Yu E, Xu W. Development and validation of a staging system for HPV-related oropharyngeal cancer by the International Collaboration on Oropharyngeal cancer Network for Staging (ICON-S): a multicentre cohort study. Lancet Oncol. 2016 Apr;17(4):440-451. doi: 10.1016/S1470-2045(15)00560-4. Epub 2016 Feb 27. PMID 26936027
- [Background] de Ruiter EJ, Ooft ML, Devriese LA, Willems SM. The prognostic role of tumor infiltrating T-lymphocytes in squamous cell carcinoma of the head and neck: A systematic review and meta-analysis. Oncoimmunology. 2017 Aug 9;6(11):e1356148. doi: 10.1080/2162402X.2017.1356148. eCollection 2017. PMID 29147608
- [Background] Hecht M, Gostian AO, Eckstein M, Rutzner S, von der Grun J, Illmer T, Hautmann MG, Klautke G, Laban S, Brunner T, Hinke A, Becker I, Frey B, Semrau S, Geppert CI, Hartmann A, Balermpas P, Budach W, Gaipl US, Iro H, Fietkau R. Safety and efficacy of single cycle induction treatment with cisplatin/docetaxel/ durvalumab/tremelimumab in locally advanced HNSCC: first results of CheckRad-CD8. J Immunother Cancer. 2020 Oct;8(2):e001378. doi: 10.1136/jitc-2020-001378. PMID 33023982
- [Background] Wondergem NE, Nauta IH, Muijlwijk T, Leemans CR, van de Ven R. The Immune Microenvironment in Head and Neck Squamous Cell Carcinoma: on Subsets and Subsites. Curr Oncol Rep. 2020 Jun 29;22(8):81. doi: 10.1007/s11912-020-00938-3. PMID 32602047
- [Background] Echarti A, Hecht M, Buttner-Herold M, Haderlein M, Hartmann A, Fietkau R, Distel L. CD8+ and Regulatory T cells Differentiate Tumor Immune Phenotypes and Predict Survival in Locally Advanced Head and Neck Cancer. Cancers (Basel). 2019 Sep 19;11(9):1398. doi: 10.3390/cancers11091398. PMID 31546872
- [Background] Rudolf J, Buttner-Herold M, Erlenbach-Wunsch K, Posselt R, Jessberger J, Haderlein M, Hecht M, Hartmann A, Fietkau R, Distel L. Regulatory T cells and cytotoxic T cells close to the epithelial-stromal interface are associated with a favorable prognosis. Oncoimmunology. 2020 Apr 14;9(1):1746149. doi: 10.1080/2162402X.2020.1746149. eCollection 2020. PMID 32363115
- [Background] Posselt R, Erlenbach-Wunsch K, Haas M, Jessberger J, Buttner-Herold M, Haderlein M, Hecht M, Hartmann A, Fietkau R, Distel LV. Spatial distribution of FoxP3+ and CD8+ tumour infiltrating T cells reflects their functional activity. Oncotarget. 2016 Sep 13;7(37):60383-60394. doi: 10.18632/oncotarget.11039. PMID 27494875
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Wimmer S, Deloch L, Hader M, Derer A, Grottker F, Weissmann T, Hecht M, Gostian AO, Fietkau R, Frey B, Gaipl US. Hypofractionated Radiotherapy Upregulates Several Immune Checkpoint Molecules in Head and Neck Squamous Cell Carcinoma Cells Independently of the HPV Status While ICOS-L Is Upregulated Only on HPV-Positive Cells. Int J Mol Sci. 2021 Aug 24;22(17):9114. doi: 10.3390/ijms22179114. PMID 34502022
- [Background] Zhou JG, Donaubauer AJ, Frey B, Becker I, Rutzner S, Eckstein M, Sun R, Ma H, Schubert P, Schweizer C, Fietkau R, Deutsch E, Gaipl U, Hecht M. Prospective development and validation of a liquid immune profile-based signature (LIPS) to predict response of patients with recurrent/metastatic cancer to immune checkpoint inhibitors. J Immunother Cancer. 2021 Feb;9(2):e001845. doi: 10.1136/jitc-2020-001845. PMID 33593828
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777
- [Background] Driehuis E, Kolders S, Spelier S, Lohmussaar K, Willems SM, Devriese LA, de Bree R, de Ruiter EJ, Korving J, Begthel H, van Es JH, Geurts V, He GW, van Jaarsveld RH, Oka R, Muraro MJ, Vivie J, Zandvliet MMJM, Hendrickx APA, Iakobachvili N, Sridevi P, Kranenburg O, van Boxtel R, Kops GJPL, Tuveson DA, Peters PJ, van Oudenaarden A, Clevers H. Oral Mucosal Organoids as a Potential Platform for Personalized Cancer Therapy. Cancer Discov. 2019 Jul;9(7):852-871. doi: 10.1158/2159-8290.CD-18-1522. Epub 2019 May 3. PMID 31053628
- [Background] Tanaka N, Osman AA, Takahashi Y, Lindemann A, Patel AA, Zhao M, Takahashi H, Myers JN. Head and neck cancer organoids established by modification of the CTOS method can be used to predict in vivo drug sensitivity. Oral Oncol. 2018 Dec;87:49-57. doi: 10.1016/j.oraloncology.2018.10.018. Epub 2018 Oct 23. PMID 30527243